CLINICAL TRIAL: NCT00254111
Title: Ultra Probe Laser System Osteoarthritis of the Hand Clinical Study.
Brief Title: Study of the Use of Laser Light to Treat Osteoarthritis of the Hand.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TriTech Manufacturing (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TT-OAV3-70505
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; hand; laser; device; hand pain; stiffness
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: Ultra Probe Laser System

SUMMARY:
The purpose of this study is to determine whether low level light therapy is effective in the treatment of osteoarthritis of the hand, when the treatment is applied to the hand by an individual in his or her own home.

DETAILED DESCRIPTION:
Osteoarthritis of the hand is a disease that breaks down the cartilage and causes formation of new bone around the joints of the hand, resulting in pain, discomfort, and often lowered ability to move the affected joints. Existing methods of treatment for osteoarthritis of the hand include oral and topical medications, physical therapy, occupational therapy, assistive device use, braces and surgery. This study is intended to evaluate the effectiveness of at-home use of a low level laser device in reducing the symptoms of osteoarthritis of the hand.

Comparison(s): Active low level laser units in addition to rescue pain medication, compared to non-active ('fake') low level laser units in addition to rescue pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiographic diagnosis of osteoarthritis of the hand.
* Hand symptoms such as pain, aching and stiffness present across the prior six months.
* Willingness to use only Tylenol to relieve hand symptoms during the study.
* Primary spoken language is English.

Exclusion Criteria:

* Current use of narcotics, opiates, morphine, steroids.
* Previous surgery to the hand.
* Infection or wound in the hand.
* Involvement in litigation, worker's compensation claim or receiving disability benefits because of osteoarthritis of the hand.
* Participation in a research study during the prior 90 days.
* Pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Study Completion 2006-07

PRIMARY OUTCOMES:
Hand pain rating on the VAS at 10 days after treatment onset.

SECONDARY OUTCOMES:
Hand pain rating on the VAS at 6 weeks after treatment onset,
Hand Range of Motion measurements at 10 days after treatment onset and at 6 weeks after treatment onset,
Rescue medication use at 10 days after treatment onset and at 6 weeks after treatment onset,
Scores on the Michigan Hand Outcomes Questionnaire at 10 days after treatment onset and at 6 weeks after treatment onset,
Study outcome satisfaction rating at 10 days after treatment onset and at 6 weeks after treatment onset,
Perceived group assignment by subjects at 10 days after treatment onset and at 6 weeks after treatment onset.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Walls, M.B.A., RAS, Study Director — Regulatory Insight, Inc.
Locations (3):
- United States (3):
  - Proctology Associates, Phoenix, Arizona
  - Advanced Wellness Center, Long Beach, California
  - Advanced Chiropractic, Bloomington, Minnesota